CLINICAL TRIAL: NCT01798849
Title: A Single Rising Dose Clinical Trial to Study the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-8892
Brief Title: A Rising Single Dose Study of the Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics of MK-8892 (MK-8892-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8892-001; 2012-005472-34 (EudraCT Number)
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-05

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Panel A-Healthy (Experimental): Within each of the 5 rising dose treatment periods, 6 participants received a single dose of MK-8892 0.5 mg, 2.0 mg, 6.0 mg, 14 mg or 2.0 mg fed, and 2 participants received placebo. Dosing periods will alternate with Panel B.
  Interventions: Drug: MK-8892; Drug: Placebo for MK-8892
- Panel B-Healthy (Experimental): Within each of the 4 rising dose treatment periods, 6 participants received a single dose of MK-8892 1.0 mg, 4.0 mg, 9.0 mg or 12 mg, and 2 participants received placebo. Dosing periods will alternate with Panel A.
  Interventions: Drug: MK-8892; Drug: Placebo for MK-8892
- Panel C-Mild/Moderate Hypertension (Experimental): Within each of the 5 single dose treatment periods, 6 participants with mild to moderate hypertension received a single dose of MK-8892 0.5 mg, 1.0 mg, 2.0 mg or 6.0 mg, and 2 participants received placebo. Dosages will be determined by the results of Panels A and B.
  Interventions: Drug: MK-8892; Drug: Placebo for MK-8892

INTERVENTIONS:
Drug: MK-8892
Drug: Placebo for MK-8892

SUMMARY:
This study will evaluate safety, tolerability and effects on central diastolic blood pressure (cDBP) of MK-8892 given as single oral doses in healthy male participants (Panel A and B) and in male participants with mild-to-moderate hypertension (Panel C).

DETAILED DESCRIPTION:
Up to three planned panels of either 8 healthy participants (Panels A and B) or 8 participants with mild to moderate hypertension (Panel C) will be enrolled. In Panels A and B, 8 participants will alternately receive single rising doses of MK-8892 or placebo. All doses will be administered in the fasted state, except Panel A, Period 5 in which a standard high-fat breakfast provided approximately 30 minutes prior to dosing.

Panel A will begin first. At least 3 days will elapse before participants in the alternate panel (Panel B) will receive the next higher dose. In Panel C, 8 mild to moderate hypertensive male participants will receive single rising doses of MK-8892 or placebo. Panel C may begin after the first 4 periods of Panels A and B have completed dosing. For all panels, there will be at least 7 days washout between treatment periods for any given participant. Participants may only be enrolled in one panel of the study. Subsequent doses in any panel will be administered only after careful evaluation of safety, tolerability, and pharmacodynamic effects of a given dose. All participants in periods of all panels (with exception of 2.0 mg fasted/fed periods) will be randomly assigned to either study drug or placebo, i.e a participant could be assigned to receive study drug in one period and placebo in another. As per the protocol allocation plan, the same participants will receive 2.0 mg MK-8892 in a fasted and fed state.The 2.0 mg MK-8892 fed/fasted data will be utilized for pharmacokinetic comparison and only the 2.0 mg MK-8892 fasted data will utilized for the analysis of the pharmacodynamics endpoints.

In addition, during any of the treatment periods if a participant demonstrates change in any one of the protocol-defined parameters lasting ≥1 hour, dose escalation in that participant will be halted and the participant may be withdrawn from the study or rechallenged at same dose or at a lower dose. Paricipants that meet criteria listed will be followed up until parameters no longer meet stopping rule criteria.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure (SBP) > 110 and ≤ 140 mmHg for Panels A and B, SBP values of 140-175 mmHg and diastolic blood pressure (DBP) of 90-105 mmHg on at least three different occasions at the prestudy (screening) visit for Panel C. Participants being treated with medication for their hypertension may be included as long as they are titrated off of their medication
* Body Mass Index (BMI) ≥ 18 kg/m^2 and ≤ 32 kg/m^2
* Healthy (with the exception of hypertensive subjects in Panel C)
* No clinically significant abnormality on electrocardiogram (ECG)
* No history of clinically significant cardiac disease
* No history of heart failure
* Nonsmoker and/or has not used nicotine or nicotine-containing products for at least 6 months

Exclusion Criteria:

* Mentally or legally incapacitated
* History of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine, gastrointestinal, cardiovascular (except mild to moderate hypertension), hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* Functional disability that can interfere with rising from a sitting position to the standing position
* History of cancer (malignancy)
* History of significant multiple and/or severe allergies (e.g. food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or food
* Positive for hepatitis B, hepatitis C, or Human Immunodeficiency Virus (HIV)
* Has had major surgery, donated or lost 1 unit of blood or participated in another investigational study within 4 weeks
* Has participated in another investigational trial within 4 weeks
* Unable to refrain from or anticipates the use of any medication during the study
* Anticipates using medication for erectile dysfunction during the study
* Uses or anticipates using organic nitrates during the study (e.g. nitroglycerin, isosorbide mononitrate, isosorbide dinitrate, pentaerythritol)
* Anticipates using cytochrome P450 inhibitors (e.g. ketoconazole) or inducers (e.g. rifampin) during the study
* Consumes excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages per day
* Consumes excessive amounts, defined as greater than 6 servings of coffee, tea, cola, or other caffeinated beverages per day
* Regular user (including recreational user) of illicit drugs or has a history of drug (including alcohol) abuse within approximately 1 year

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-03-15 (Actual); Primary Completion 2013-07-17 (Actual); Study Completion 2013-07-17 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Panels A and B, 8 healthy male participants alternately received single rising doses of MK-8892 or placebo.In Panel C, 8 mild to moderate hypertensive male participants received single rising doses of MK-8892 determined by results of Panels A and B or placebo. Each period in a panel was separated by a 7-day washout.
Groups:
- Panel A-Healthy: Within each of the 5 rising dose treatment periods, 6 participants received a single dose of MK-8892 0.5 mg, 2.0 mg, 6.0 mg, or 14 mg, and 2 participants received placebo. Dosing periods alternated with Panel B.
- Panel B-Healthy: Within each of the 4 rising dose treatment periods, 6 participants received a single dose of MK-8892 1.0 mg, 4.0 mg, 9.0 mg or 12 mg, and 2 participants received placebo. Dosing periods alternated with Panel A.
- Panel C-Mild/Moderate Hypertension: Within each of the 5 single dose treatment periods, 6 participants with mild to moderate hypertension received a single dose of MK-8892 0.5 mg, 1.0 mg, 2.0 mg or 6.0 mg, and 2 participants received placebo. Dosages were determined by the results of Panels A and B.
Period: Overall Study
Arm/Group | Panel A-Healthy | Panel B-Healthy | Panel C-Mild/Moderate Hypertension
Started | 8 | 8 | 9 (1 participant discontinued after Period 1 and was replaced for Periods 2-4)
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A-Healthy | Panel B-Healthy | Panel C-Mild/Moderate Hypertension | Total
Number analyzed (Participants) | 8 | 8 | 9 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (9.5) | 37.1 (15.1) | 50.6 (5.3) | 43.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 8 | 8 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Report 1 or More Adverse Events (AEs)- Healthy Participants
Description: An AE was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, regardless of whether or not it was considered related to the medicinal product. The percentage of participants that reported at least 1 AE was summarized. Adverse events were summarized by dose taken at the time of the event.
Time Frame: up to 7 weeks
Population: All healthy participants (Panels A and B) who received at least 1 dose of the study drug. As pre-specified in the protocol, safety data were pooled for the MK 8892 2.0 mg fed and fasted arms only and were not planned to be provided separately.
Measure: Number; unit: Percentage of Participants
Groups:
- 0.5 mg MK-8892-Healthy: Single oral dose of 0.5 mg MK-8892
- 1.0 mg MK-8892-Healthy: Single oral dose of 1.0 mg MK-8892
- 2.0 mg MK-8892-Healthy (Pooled): Single oral dose of 2.0 mg MK-8892
- 4.0 mg MK-8892-Healthy: Single oral dose of 4.0 mg MK-8892
- 6.0 mg MK-8892-Healthy: Single oral dose of 6.0 mg MK-8892
- 9.0 mg MK-8892-Healthy: Single oral dose of 9.0 mg MK-8892
- 12.0 mg MK-8892-Healthy: Single oral dose of 12.0 mg MK-8892
- 14.0 mg MK-8892-Healthy: Single oral dose of 14.0 mg MK-8892
- Placebo-Healthy: Single oral dose of placebo to match MK-8892
Arm/Group | 0.5 mg MK-8892-Healthy | 1.0 mg MK-8892-Healthy | 2.0 mg MK-8892-Healthy (Pooled) | 4.0 mg MK-8892-Healthy | 6.0 mg MK-8892-Healthy | 9.0 mg MK-8892-Healthy | 12.0 mg MK-8892-Healthy | 14.0 mg MK-8892-Healthy | Placebo-Healthy
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Percentage of Participants | 50.0 | 66.7 | 50.0 | 100.0 | 100.0 | 83.3 | 100.0 | 100.0 | 43.8

2. Primary Outcome: Percentage of Participants Who Were Discontinued From the Study Due to an AE- Healthy Participants
Description: An AE was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, regardless of whether or not considered related to the medicinal product. The percentage of participants that were discontinued from the study due to an AE was summarized. Adverse events were summarized by dose taken at the time of the event.
Time Frame: up to 7 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 0.5 mg MK-8892-Healthy | 1.0 mg MK-8892-Healthy | 2.0 mg MK-8892-Healthy (Pooled) | 4.0 mg MK-8892-Healthy | 6.0 mg MK-8892-Healthy | 9.0 mg MK-8892-Healthy | 12.0 mg MK-8892-Healthy | 14.0 mg MK-8892-Healthy | Placebo-Healthy
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

3. Primary Outcome: Change in 24-hour Time-weighted Average (TWA0-24hr) for Central Diastolic Blood Pressure (cDBP)- Healthy Participants
Description: Central diastolic blood pressure measurements were obtained at predose and at 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose via applanation tonometry of the radial artery. The average central diastolic blood pressure over the 24-hour monitoring period was calculated for each dose of each panel by adjusting each time-point by the baseline, aggregating the area under the curve (AUC) by the trapezoidal method and then dividing the AUC by 24 hours. A negative number indicates a decrease.
Time Frame: Predose (baseline) and 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose (for each Dosing Period of Each Panel)
Population: Healthy participants (Panels A and B) who were administered study drug in a fasted state, who complied with the protocol sufficiently to ensure that these data were likely to exhibit the effects of the treatment, according to the underlying scientific model and had data available for endpoint.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- 2.0 mg MK-8892-Healthy: Single oral dose of 2.0 mg MK-8892
Arm/Group | 0.5 mg MK-8892-Healthy | 1.0 mg MK-8892-Healthy | 2.0 mg MK-8892-Healthy | 4.0 mg MK-8892-Healthy | 6.0 mg MK-8892-Healthy | 9.0 mg MK-8892-Healthy | 12.0 mg MK-8892-Healthy | 14.0 mg MK-8892-Healthy | Placebo-Healthy
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
mm Hg | -1.83 (1.71) | -2.27 (1.69) | -4.21 (1.70) | -4.25 (1.71) | -6.22 (1.70) | -6.64 (1.69) | -6.94 (1.69) | -8.89 (1.70) | -1.33 (1.26)
Statistical Analysis 1: Comparison: 0.5 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.732, Mixed effect model; Mixed effects model for each cohort containing fixed effects for Day 1 predose and treatment and a random effect for participant; Difference in Least-square (LS) Means = -0.50, 95% CI 2-sided [-3.42 to 2.43] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 2: Comparison: 1.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.531, Mixed effects model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -0.94, 95% CI 2-sided [-3.94 to 2.06] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 3: Comparison: 2.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.056, Mixed effects model; [statistical method as in outcome 3, analysis 1]; Difference in LS Means = -2.88, 95% CI 2-sided [-5.83 to 0.08] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 4: Comparison: 4.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.063, Mixed effects model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -2.92, 95% CI 2-sided [-6.00 to 0.17] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 5: Comparison: 6.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.002, Mixed effects model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -4.89, 95% CI 2-sided [-7.79 to -1.99] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 6: Comparison: 9.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.001, Mixed effects model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -5.31, 95% CI 2-sided [-8.32 to -2.31] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 7: Comparison: 12.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.001, Mixed effects model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -5.61, 95% CI 2-sided [-8.62 to -2.60] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 8: Comparison: 14.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p < 0.0001, Mixed effects model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -7.56, 95% CI 2-sided [-10.50 to -4.63] — Difference in LS means = LS mean MK-8892 minus LS mean placebo

4. Primary Outcome: Percentage of Participants Who Report 1 or More Adverse Events (AEs) - Hypertensive Participants
Description: An AE was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. The percentage of participants that reported at least 1 AE was summarized. Adverse events were summarized by dose taken at the time of the event.
Time Frame: up to 7 weeks
Population: All hypertensive participants (Panel C) who received at least 1 dose of the study drug in a fasted state.
Measure: Number; unit: Percentage of Participants
Groups:
- 0.5 mg MK-8892-Hypertensive: Single oral dose of 0.5 mg MK-8892
- 1.0 mg MK-8892-Hypertensive: Single oral dose of 1.0 mg MK-8892
- 2.0 mg MK-8892-Hypertensive: single oral dose of 2.0 mg MK-8892
- 6.0 mg MK-8892-Hypertensive: Single oral dose of 6.0 mg MK-8892. Includes rechallenge
- Placebo-Hypertensive: Single oral dose of placebo to match MK-8892
Arm/Group | 0.5 mg MK-8892-Hypertensive | 1.0 mg MK-8892-Hypertensive | 2.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive | Placebo-Hypertensive
Number analyzed (Participants) | 6 | 6 | 6 | 9 | 8
Percentage of Participants | 50.0 | 33.3 | 66.7 | 77.8 | 75.0

5. Primary Outcome: Percentage of Participants Who Were Discontinued From the Due to an AE - Hypertensive Participants
Description: An AE was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. The percentage of participants that were discontinued from the study due to an AE was summarized. Adverse events were summarized by dose taken at the time of the event.
Time Frame: up to 7 weeks
Population: All hypertensive participants (Panel C) who received at least 1 dose of the study drug in a fasted state.
Measure: Number; unit: Percentage of Participants
Arm/Group | 0.5 mg MK-8892-Hypertensive | 1.0 mg MK-8892-Hypertensive | 2.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive | Placebo-Hypertensive
Number analyzed (Participants) | 6 | 6 | 6 | 9 | 8
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

6. Primary Outcome: Change in 24-hour Time-weighted Average (TWA0-24hr) for Central Diastolic Blood Pressure (cDBP) - Hypertensive Participants
Description: Central diastolic blood pressure measurements were obtained at predose and 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose via applanation tonometry of the radial artery. The average central diastolic blood pressure over the 24-hour monitoring period was calculated for each dose of each panel by adjusting each time-point by the baseline, aggregating the area under the curve (AUC) by the trapezoidal method and then dividing the AUC by 24 hours. A negative number indicates a decrease.
Time Frame: Predose (baseline) and 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose (for each Dosing Period)
Population: Hypertensive participants (Panel C) who were administered study drug in a fasted state, who complied with the protocol sufficiently to ensure that these data were likely to exhibit the effects of the treatment, according to the underlying scientific model and had data available for endpoint.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- 6.0 mg MK-8892-Hypertensive: Single oral dose of 6.0 mg MK-8892
Arm/Group | 0.5 mg MK-8892-Hypertensive | 1.0 mg MK-8892-Hypertensive | 2.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive | Placebo-Hypertensive
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
mm Hg | -3.56 (1.87) | -4.76 (1.85) | -7.55 (1.85) | -7.86 (1.59) | -1.22 (1.67)
Statistical Analysis 1: Comparison: 0.5 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p = 0.165, Mixed effects model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -2.34, 95% CI 2-sided [-5.70 to 1.02] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 2: Comparison: 1.0 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p = 0.038, Mixed effects model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -3.53, 95% CI 2-sided [-6.86 to -0.21] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 3: Comparison: 2.0 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p = 0.000, Mixed effects model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -6.32, 95% CI 2-sided [-9.55 to -3.10] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 4: Comparison: 6.0 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p < 0.0001, Mixed effects model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -6.63, 95% CI 2-sided [-9.35 to -3.92] — Difference in LS means = LS mean MK-8892 minus LS mean placebo

7. Secondary Outcome: Change in TWA0-24hrs for Peripheral Diastolic Blood Pressure (pDBP) - Healthy Participants
Description: Peripheral diastolic blood pressure was measured using a validated automatic measuring device. The time-weighted average change from baseline was calculated by adjusting each time-point by the baseline, aggregating the area under the curve (AUC) by the trapezoidal method and then dividing the AUC by 24 hours. A negative number indicates a decrease.
Time Frame: Predose and 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose (for each Dosing Period of Each Panel)
Population: Healthy participants (Panels and B) who were administered study drug in a fasted state, who complied with the protocol sufficiently to ensure that these data were likely to exhibit the effects of the treatment, according to the underlying scientific model and had data available for endpoint.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | 0.5 mg MK-8892-Healthy | 1.0 mg MK-8892-Healthy | 2.0 mg MK-8892-Healthy | 4.0 mg MK-8892-Healthy | 6.0 mg MK-8892-Healthy | 9.0 mg MK-8892-Healthy | 12.0 mg MK-8892-Healthy | 14.0 mg MK-8892-Healthy | Placebo-Healthy
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
mm Hg | -4.34 (1.73) | -2.43 (0.83) | -3.69 (1.10) | -4.50 (1.49) | -6.56 (1.06) | -7.04 (0.99) | -7.35 (0.71) | -9.89 (1.68) | -1.67 (0.82)
Statistical Analysis 1: Comparison: 0.5 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.128, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -2.67, 95% CI 2-sided [-6.14 to 0.80] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 2: Comparison: 1.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.305, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -0.76, 95% CI 2-sided [-2.24 to 0.72] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 3: Comparison: 2.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.070, Mixed effects model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -2.03, 95% CI 2-sided [-4.23 to 0.17] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 4: Comparison: 4.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.036, Mixed effects model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -2.84, 95% CI 2-sided [-5.48 to -0.19] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 5: Comparison: 6.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p < 0.0001, Mixed effects model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -4.89, 95% CI 2-sided [-6.40 to -3.37] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 6: Comparison: 9.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p < 0.0001, Mixed effects model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -5.37, 95% CI 2-sided [-7.29 to -3.46] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 7: Comparison: 12.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p < 0.0001, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -5.68, 95% CI 2-sided [-6.70 to -4.65] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 8: Comparison: 14.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p < 0.0001, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -8.22, 95% CI 2-sided [-11.95 to -4.50] — Difference in LS means = LS mean MK-8892 minus LS mean placebo

8. Secondary Outcome: Change in TWA0-24hrs for Heart Rate (HR) - Healthy Participants
Description: Heart rate was measured predose and every 30 minutes from 0.5-4 hours postdose; hourly from 4-12 hours postdose; every 2 hours from 12-16 hours postdose; and at 24 postdose by a validated automatic measuring device. The time-weighted average change from baseline was calculated by adjusting each time-point by the baseline, aggregating the area under the curve (AUC) by the trapezoidal method and then dividing the AUC by 24 hours. A negative number indicates a decrease.
Time Frame: Predose (baseline) and every 30 minutes from 0.5-4 hours postdose; hourly from 4-12 hours postdose; every 2 hours from 12-16 hours postdose; and at 24 postdose (for each Dosing Period of Each Panel)
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 0.5 mg MK-8892-Healthy | 1.0 mg MK-8892-Healthy | 2.0 mg MK-8892-Healthy | 4.0 mg MK-8892-Healthy | 6.0 mg MK-8892-Healthy | 9.0 mg MK-8892-Healthy | 12.0 mg MK-8892-Healthy | 14.0 mg MK-8892-Healthy | Placebo-Healthy
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
beats per minute (bpm) | 0.46 (1.36) | 5.55 (1.32) | 4.71 (1.42) | 7.44 (1.93) | 9.29 (2.22) | 8.85 (1.93) | 10.34 (1.09) | 16.29 (2.21) | 2.23 (1.11)
Statistical Analysis 1: Comparison: 0.5 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.212, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -1.77, 95% CI 2-sided [-4.59 to 1.05] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 2: Comparison: 1.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.050, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = 3.32, 95% CI 2-sided [0.00 to 6.64] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 3: Comparison: 2.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.016, Mixed effect model; Difference in LS means = 2.48, 95% CI 2-sided [0.49 to 4.47] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 4: Comparison: 4.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.007, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = 5.21, 95% CI 2-sided [1.51 to 8.92] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 5: Comparison: 6.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.001, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = 7.06, 95% CI 2-sided [3.03 to 11.10] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 6: Comparison: 9.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.002, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = 6.62, 95% CI 2-sided [2.54 to 10.71] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 7: Comparison: 12.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p < 0.0001, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = 8.11, 95% CI 2-sided [5.45 to 10.76] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 8: Comparison: 14.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p < 0.0001, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = 14.05, 95% CI 2-sided [10.54 to 17.57] — Difference in LS means = LS mean MK-8892 minus LS mean placebo

9. Secondary Outcome: Change in TWA0-24hr for Augmentation Index (AIx) - Healthy Participants
Description: AIx was measured by applanation tonometry of the radial artery. The central pressure waveform was determined from the peripheral pressure waveform by a transfer function. Augmentation index is the percentage of the central pulse pressure attributed to the reflected pulse wave, and is an indirect measure of systemic arterial stiffness. The time-weighted average change from baseline was calculated by adjusting each time-point by the baseline, aggregating the area under the curve (AUC) by the trapezoidal method and then dividing the AUC by 24 hours.
Time Frame: Predose (baseline) and 2, 4, 12, and 24 hours postdose (for each Dosing Period of Each Panel)
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | 0.5 mg MK-8892-Healthy | 1.0 mg MK-8892-Healthy | 2.0 mg MK-8892-Healthy | 4.0 mg MK-8892-Healthy | 6.0 mg MK-8892-Healthy | 9.0 mg MK-8892-Healthy | 12.0 mg MK-8892-Healthy | 14.0 mg MK-8892-Healthy | Placebo-Healthy
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Percentage | -1.73 (2.30) | -2.31 (2.32) | -2.82 (2.31) | -0.26 (2.38) | -4.23 (2.29) | -3.85 (2.31) | -1.84 (2.30) | -4.81 (2.32) | -0.07 (2.06)
Statistical Analysis 1: Comparison: 0.5 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.202, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -1.66, 95% CI 2-sided [-4.24 to 0.93] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 2: Comparison: 1.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.115, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -2.23, 95% CI 2-sided [-5.03 to 0.57] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 3: Comparison: 2.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.043, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -2.75, 95% CI 2-sided [-5.40 to -0.09] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 4: Comparison: 4.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.901, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -0.19, 95% CI 2-sided [-3.22 to 2.84] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 5: Comparison: 6.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.002, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Mixed effect model = -4.15, 95% CI 2-sided [-6.74 to -1.57] — Mixed effects model for each cohort containing fixed effects for Day 1 predose and treatment and a random effect for participant
Statistical Analysis 6: Comparison: 9.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.008, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -3.77, 95% CI 2-sided [-6.48 to -1.06] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 7: Comparison: 12.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.201, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -1.77, 95% CI 2-sided [-4.51 to 0.98] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 8: Comparison: 14.0 mg MK-8892-Healthy vs Placebo-Healthy; Test type: Other; p = 0.001, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -4.74, 95% CI 2-sided [-7.37 to -2.11] — Difference in LS means = LS mean MK-8892 minus LS mean placebo

10. Secondary Outcome: Change in TWA0-24hrs for Peripheral Diastolic Blood Pressure (pDBP) - Hypertensive Participants
Description: Peripheral blood pressure assessments were obtained at predose and 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose by using a validated automatic measuring device. Peripheral diastolic blood pressure was measured a validated automatic measuring device. The time-weighted average change from baseline was calculated by adjusting each time-point by the baseline, aggregating the area under the curve (AUC) by the trapezoidal method and then dividing the AUC by 24 hours. Negative number indicates a decrease.
Time Frame: Predose (baseline) and 2, 3, 4, 6, 8, 12, 16 and 24 hours postdose (for each Dosing Period of Each Panel)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | 0.5 mg MK-8892-Hypertensive | 1.0 mg MK-8892-Hypertensive | 2.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive | Placebo-Hypertensive
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
mm Hg | -3.40 (1.13) | -4.17 (1.63) | -7.29 (1.40) | -9.16 (1.43) | -0.87 (1.40)
Statistical Analysis 1: Comparison: 0.5 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p = 0.042, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -2.53, 95% CI 2-sided [-4.97 to -0.10] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 2: Comparison: 1.0 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p = 0.010, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -3.29, 95% CI 2-sided [-5.71 to -0.88] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 3: Comparison: 2.0 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p < 0.0001, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -6.42, 95% CI 2-sided [-8.94 to -3.89] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 4: Comparison: 6.0 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p < 0.0001, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -8.28, 95% CI 2-sided [-11.32 to -5.25] — Difference in LS means = LS mean MK-8892 minus LS mean placebo

11. Secondary Outcome: Change in TWA0-24hrs for Heart Rate (HR) - Hypertensive Participants
Description: Heart rate was measured predose and every 30 minutes from 0.5-4 hours postdose; hourly from 4-12 hours postdose; every 2 hours from 12-16 hours postdose; and at 24 postdose by a validated automatic measuring device. The time-weighted average change from baseline was calculated by adjusting each time-point by the baseline, aggregating the area under the curve (AUC) by the trapezoidal method and then dividing the AUC by 24 hours. Negative number indicates a decrease.
Time Frame: Predose and every 30 minutes from 0.5-4 hours postdose; hourly from 4-12 hours postdose; every 2 hours from 12-16 hours postdose; and at 24 postdose (for each Dosing Period of Each Panel)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | 0.5 mg MK-8892-Hypertensive | 1.0 mg MK-8892-Hypertensive | 2.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive | Placebo-Hypertensive
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
bpm | -0.92 (1.59) | -0.74 (1.88) | 0.87 (1.92) | 7.68 (1.51) | -1.46 (1.62)
Statistical Analysis 1: Comparison: 0.5 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p = 0.638, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = 0.54, 95% CI 2-sided [-1.80 to 2.87] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 2: Comparison: 1.0 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p = 0.616, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = 0.72, 95% CI 2-sided [-2.20 to 3.63] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 3: Comparison: 2.0 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p = 0.041, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = 2.33, 95% CI 2-sided [0.11 to 4.56] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 4: Comparison: 6.0 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p < 0.0001, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = 9.14, 95% CI 2-sided [6.98 to 11.30] — Difference in LS means = LS mean MK-8892 minus LS mean placebo

12. Secondary Outcome: TWA0-24hr for Augmentation Index (AIx) - Hypertensive Participants
Description: AIx was measured by applanation tonometry of the radial artery. The central pressure waveform was determined from the peripheral pressure waveform by a transfer function. Augmentation index is the percentage of the central pulse pressure attributed to the reflected pulse wave, and is an indirect measure of systemic arterial stiffness. The time-weighted average change from baseline was calculated by adjusting each time-point by the baseline, aggregating the area under the curve (AUC) by the trapezoidal method and then dividing the AUC by 24 hours. Negative number indicates a decrease.
Time Frame: Predose to 24 hours Postdose (for each Dosing Period of Each Panel)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | 0.5 mg MK-8892-Hypertensive | 1.0 mg MK-8892-Hypertensive | 2.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive | Placebo-Hypertensive
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Percentage | -2.30 (2.01) | -2.57 (2.01) | -3.94 (2.01) | -5.43 (1.80) | -1.65 (1.86)
Statistical Analysis 1: Comparison: 0.5 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p = 0.677, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -0.65, 95% CI 2-sided [-3.81 to 2.52] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 2: Comparison: 1.0 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p = 0.554, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -0.92, 95% CI 2-sided [-4.08 to 2.24] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 3: Comparison: 2.0 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p = 0.137, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -2.29, 95% CI 2-sided [-5.35 to 0.78] — Difference in LS means = LS mean MK-8892 minus LS mean placebo
Statistical Analysis 4: Comparison: 6.0 mg MK-8892-Hypertensive vs Placebo-Hypertensive; Test type: Other; p = 0.006, Mixed effect model; [statistical method as in outcome 3, analysis 1]; Difference in LS means = -3.78, 95% CI 2-sided [-6.37 to -1.19] — Difference in LS means = LS mean MK-8892 minus LS mean placebo

13. Secondary Outcome: Area Under the Concentration Time-curve From Hour 0 to 24 Hours (AUC0-24hr) of MK-8892 - Healthy Participants
Description: Blood samples taken at Predose, 0.5, 1, 2, 4, 6, 8, 12, 16, and 24 hours postdose of each dosing period to determine the AUC0-24hr.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8, 12, 16, and 24 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM·hr
Arm/Group | 0.5 mg MK-8892-Healthy | 1.0 mg MK-8892-Healthy | 2.0 mg MK-8892-Healthy | 4.0 mg MK-8892-Healthy | 6.0 mg MK-8892-Healthy | 9.0 mg MK-8892-Healthy | 12.0 mg MK-8892-Healthy | 14.0 mg MK-8892-Healthy
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 5
nM·hr | 67 (27) | 128 (32) | 218 (11) | 464 (28) | 694 (14) | 793 (31) | 1202 (25) | 1306 (18)

14. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Measurable Plasma Concentration Time Point (AUC0-last) of MK-8892 - Healthy Participants
Description: Blood samples taken at Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose of each dosing period to determine the AUC0-last.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM·hr
Arm/Group | 0.5 mg MK-8892-Healthy | 1.0 mg MK-8892-Healthy | 2.0 mg MK-8892-Healthy | 4.0 mg MK-8892-Healthy | 6.0 mg MK-8892-Healthy | 9.0 mg MK-8892-Healthy | 12.0 mg MK-8892-Healthy | 14.0 mg MK-8892-Healthy
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 5
nM·hr | 103.3 (40.0) | 216.8 (58.7) | 368.5 (29.2) | 724.7 (42.9) | 1157.6 (26.4) | 1293.3 (39.4) | 2286.3 (35.7) | 2527.7 (25.5)

15. Secondary Outcome: Area Under the Concentration Time-curve From Hour 0 to Infinity (AUC0-inf) of MK-8892 - Healthy Participants
Description: Blood samples taken at Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose of each dosing period to determine the AUC0-inf.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM·hr
Arm/Group | 0.5 mg MK-8892-Healthy | 1.0 mg MK-8892-Healthy | 2.0 mg MK-8892-Healthy | 4.0 mg MK-8892-Healthy | 6.0 mg MK-8892-Healthy | 9.0 mg MK-8892-Healthy | 12.0 mg MK-8892-Healthy | 14.0 mg MK-8892-Healthy
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 5
nM·hr | 113 (37) | 232 (63) | 391 (34) | 757 (50) | 1195 (30) | 1342 (41) | 2443 (39) | 2702 (31)

16. Secondary Outcome: Maximum Concentration (Cmax) of MK-8892 - Healthy Participants
Description: Blood samples taken at Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose of each dosing period to determine the Cmax.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | 0.5 mg MK-8892-Healthy | 1.0 mg MK-8892-Healthy | 2.0 mg MK-8892-Healthy | 4.0 mg MK-8892-Healthy | 6.0 mg MK-8892-Healthy | 9.0 mg MK-8892-Healthy | 12.0 mg MK-8892-Healthy | 14.0 mg MK-8892-Healthy
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 5
nM | 4.8 (32) | 8.5 (23) | 17.9 (19) | 35.6 (26) | 49.0 (21) | 52.8 (38) | 72.8 (23) | 87.3 (16)

17. Secondary Outcome: Time to Cmax (Tmax) of MK-8892 - Healthy Participants
Description: Blood samples taken at Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose of each dosing period to determine the Tmax.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | 0.5 mg MK-8892-Healthy | 1.0 mg MK-8892-Healthy | 2.0 mg MK-8892-Healthy | 4.0 mg MK-8892-Healthy | 6.0 mg MK-8892-Healthy | 9.0 mg MK-8892-Healthy | 12.0 mg MK-8892-Healthy | 14.0 mg MK-8892-Healthy
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 5
hours | 4 [2 to 6] | 4 [1 to 6] | 4 [1 to 6] | 4 [1 to 6] | 4 [2 to 6] | 5 [4 to 8] | 4 [4 to 8] | 2 [1 to 8]

18. Secondary Outcome: Apparent Terminal Half-life (t1/2) of MK-8892 - Healthy Participants
Description: Blood samples taken at Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose of each dosing period to determine the t1/2.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 0.5 mg MK-8892-Healthy | 1.0 mg MK-8892-Healthy | 2.0 mg MK-8892-Healthy | 4.0 mg MK-8892-Healthy | 6.0 mg MK-8892-Healthy | 9.0 mg MK-8892-Healthy | 12.0 mg MK-8892-Healthy | 14.0 mg MK-8892-Healthy
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 5
Hours | 17.9 (28) | 20.6 (40) | 20.1 (44) | 17.7 (43) | 15.6 (45) | 20.9 (28) | 23.7 (23) | 21.1 (41)

19. Secondary Outcome: Area Under the Concentration Time-curve From Hour 0 to 24 Hours (AUC0-24hr) of MK-8892 - Hypertensive Participants
Description: Blood samples taken at Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, and 24 hours postdose of each dosing period to determine the AUC0-24hr.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, and 24 hours postdose
Population: Hypertensive participants (Panel C) who were administered study drug in a fasted state, who complied with the protocol sufficiently to ensure that these data were likely to exhibit the effects of the treatment, according to the underlying scientific model and had data available for endpoint. Includes protocol-defined 6.0 mg rechallenge.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM·hr
Groups:
- 6.0 mg MK-8892-Hypertensive - Rechallenge: Participants who were assigned to 6.0 mg HT group who were administered a rechallenge 6.0 mg dose of MK-8892
Arm/Group | 0.5 mg MK-8892-Hypertensive | 1.0 mg MK-8892-Hypertensive | 2.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive - Rechallenge
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
nM·hr | 79 (27) | 158 (14) | 285 (17) | 806 (24) | 714 (22)

20. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Measurable Plasma Concentration Time Point (AUC0-last) of MK-8892 - Hypertensive Participants
Description: as for outcome 14
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose
Population: Hypertensive participants (Panel C) who complied with the protocol sufficiently to ensure that these data were likely to exhibit the effects of the treatment, according to the underlying scientific model and had data available for endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM·hr
Arm/Group | 0.5 mg MK-8892-Hypertensive | 1.0 mg MK-8892-Hypertensive | 2.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive - Rechallenge
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
nM·hr | 150.2 (45.9) | 317.3 (25.9) | 522.3 (24.0) | 1700.2 (38.5) | 1538.8 (23.5)

21. Secondary Outcome: Area Under the Concentration Time-curve From Hour 0 to Infinity (AUC0-inf) of MK-8892- Hypertensive Participants
Description: as for outcome 15
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM·hr
Arm/Group | 0.5 mg MK-8892-Hypertensive | 1.0 mg MK-8892-Hypertensive | 2.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive - Rechallenge
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
nM·hr | 164.0 (53.0) | 346.0 (32.0) | 557.0 (28.0) | 1947.0 (48.0) | 1760.0 (38.0)

22. Secondary Outcome: Maximum Concentration (Cmax) of MK-8892- Hypertensive Participants
Description: as for outcome 16
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | 0.5 mg MK-8892-Hypertensive | 1.0 mg MK-8892-Hypertensive | 2.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive - Rechallenge
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
nM | 4.9 (21.0) | 9.8 (13.0) | 17.6 (30.0) | 48.9 (15.0) | 47.1 (33.0)

23. Secondary Outcome: Time to Cmax (Tmax) of MK-8892- Hypertensive Participants
Description: as for outcome 17
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose
Population: as for outcome 19
Measure: Median (Full Range); unit: Hours
Arm/Group | 0.5 mg MK-8892-Hypertensive | 1.0 mg MK-8892-Hypertensive | 2.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive - Rechallenge
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
Hours | 3 [1 to 6] | 4 [2 to 8] | 6 [4 to 12] | 4 [2 to 12] | 4 [4 to 8]

24. Secondary Outcome: Apparent Terminal Half-life (t1/2) of MK-8892- Hypertensive Participants
Description: as for outcome 18
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 0.5 mg MK-8892-Hypertensive | 1.0 mg MK-8892-Hypertensive | 2.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive - Rechallenge
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
Hours | 23.5 (30) | 24.5 (28) | 21.6 (34) | 28.8 (49) | 26.3 (57)

25. Secondary Outcome: Area Under the Concentration Time-curve From Hour 0 to 24 Hours (AUC0-24hr) of 2.0 mg MK-8892-Healthy Participants-Fasted/Fed
Description: Blood samples taken at Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, and 24 hours postdose of each dosing period to determine the AUC0-24hr. A mixed effects model with Cohort (Healthy or hypertensive) as a fixed term, participant as a random effect was used for summary data. For participants that participated in Period 5, study drug was administered after a standard high-fat breakfast provided approximately 30 minutes prior to dosing. The meal was consumed in a 20-minute period with start and stop times being recorded. Participants were administered a single dose of MK-8892 or matching placebo Within 10 minutes of completing the meal.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, and 24 hours postdose
Population: Healthy participants (Panel A) who were administered 2.0 mg MK-8892 in both fasted and fed state, who complied with the protocol sufficiently to ensure that these data were likely to exhibit the effects of the treatment, according to the underlying scientific model and had data available for endpoint.
Measure: Geometric Mean (90% Confidence Interval); unit: nM·hr
Groups:
- 2.0 mg MK-8892-Healthy-Fasted: Single oral dose of 2.0 mg MK-8892 after an 8-hour fast
- 2.0 mg MK-8892-Healthy-Fed: Single oral dose of 2.0 mg MK-8892 after a high-fat breakfest
Arm/Group | 2.0 mg MK-8892-Healthy-Fasted | 2.0 mg MK-8892-Healthy-Fed
Number analyzed (Participants) | 6 | 6
nM·hr | 218.2 [199.3 to 238.9] | 278.2 [241.5 to 320.4]

26. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Measurable Plasma Concentration Time Point (AUC0-last) of 2.0 mg MK-8892 - Healthy Participants-Fasted/Fed
Description: Blood samples taken at Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose of each dosing period to determine the AUC0-last. A mixed effects model with Cohort (Healthy or hypertensive) as a fixed term, participant as a random effect was used for summary data. For participants that participated in Period 5, study drug was administered after a standard high-fat breakfast provided approximately 30 minutes prior to dosing. The meal was consumed in a 20-minute period with start and stop times being recorded. Participants were administered a single dose of MK-8892 or matching placebo Within 10 minutes of completing the meal.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM·hr
Arm/Group | 2.0 mg MK-8892-Healthy-Fasted | 2.0 mg MK-8892-Healthy-Fed
Number analyzed (Participants) | 6 | 6
nM·hr | 368.5 (29.2) | 494.6 (29.2)

27. Secondary Outcome: Area Under the Concentration Time-curve From Hour 0 to Infinity (AUC0-inf) of 2.0 mg MK-8892 - Healthy Participants-Fasted/Fed
Description: Blood samples taken at Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose of each dosing period to determine the AUC0-inf. A mixed effects model with Cohort (Healthy or hypertensive) as a fixed term, participant as a random effect was used for summary data. For participants that participated in Period 5, study drug was administered after a standard high-fat breakfast provided approximately 30 minutes prior to dosing. The meal was consumed in a 20-minute period with start and stop times being recorded. Participants were administered a single dose of MK-8892 or matching placebo Within 10 minutes of completing the meal.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose
Population: as for outcome 25
Measure: Geometric Mean (90% Confidence Interval); unit: nM·hr
Arm/Group | 2.0 mg MK-8892-Healthy-Fasted | 2.0 mg MK-8892-Healthy-Fed
Number analyzed (Participants) | 6 | 6
nM·hr | 390.0 [298.7 to 509.1] | 518.5 [400.6 to 671.1]

28. Secondary Outcome: Maximum Concentration (Cmax) of 2.0 mg MK-8892 - Healthy Participants- Fasted/Fed
Description: Blood samples taken at Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose of each dosing period to determine the Cmax. A mixed effects model with Cohort (Healthy or hypertensive) as a fixed term, participant as a random effect was used for summary data. For participants that participated in Period 5, study drug was administered after a standard high-fat breakfast provided approximately 30 minutes prior to dosing. The meal was consumed in a 20-minute period with start and stop times being recorded. Participants were administered a single dose of MK-8892 or matching placebo Within 10 minutes of completing the meal.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose
Population: as for outcome 25
Measure: Geometric Mean (90% Confidence Interval); unit: nM
Arm/Group | 2.0 mg MK-8892-Healthy-Fasted | 2.0 mg MK-8892-Healthy-Fed
Number analyzed (Participants) | 6 | 6
nM | 17.9 [15.3 to 20.9] | 20.5 [17.8 to 23.6]

29. Secondary Outcome: Apparent Terminal Half-life (t1/2) of 2.0 mg MK-8892 - Healthy Participants -Fasted/Fed
Description: Blood samples taken at Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose of each dosing period to determine the t1/2.A mixed effects model with Cohort (Healthy or hypertensive) as a fixed term, participant as a random effect was used for summary data. For participants that participated in Period 5, study drug was administered after a standard high-fat breakfast provided approximately 30 minutes prior to dosing. The meal was consumed in a 20-minute period with start and stop times being recorded. Participants were administered a single dose of MK-8892 or matching placebo Within 10 minutes of completing the meal.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose
Population: as for outcome 25
Measure: Geometric Mean (90% Confidence Interval); unit: Hours
Groups:
- 2.0 mg MK-8892-Healthy -Fasted: Single oral dose of 2.0 mg MK-8892 after an 8-hour fast
- 2.0 Mg MK-8892- Healthy - Fed: single oral dose of 2.0 mg MK-8892 after a high-fat breakfest
Arm/Group | 2.0 mg MK-8892-Healthy -Fasted | 2.0 Mg MK-8892- Healthy - Fed
Number analyzed (Participants) | 6 | 6
Hours | 20.1 [14.3 to 28.5] | 20.5 [17.3 to 24.2]

ADVERSE EVENTS:
Time Frame: up to 7 weeks
Description: All participants who received at least 1 dose of the study drug. Adverse events are reported by dose taken at time of event and not by panel or sequence. As pre-specified in the protocol, safety data were pooled for the MK 8892 2.0 mg fed and fasted arms only and were not planned to be provided separately.
Arm/Group | 0.5 mg MK-8892-Healthy | 1.0 mg MK-8892-Healthy | 2.0 mg MK-8892-Healthy (Pooled) | 4.0 mg MK-8892-Healthy | 6.0 mg MK-8892-Healthy | 9.0 mg MK-8892-Healthy | 12.0 mg MK-8892-Healthy | 14.0 mg MK-8892-Healthy | Placebo-Healthy | 0.5 mg MK-8892-Hypertensive | 1.0 mg MK-8892-Hypertensive | 2.0 mg MK-8892-Hypertensive | 6.0 mg MK-8892-Hypertensive | Placebo-Hypertensive
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/16 | 0/6 | 0/6 | 0/6 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/16 | 0/6 | 0/6 | 0/6 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 3/6 | 4/6 | 3/6 | 6/6 | 6/6 | 5/6 | 6/6 | 6/6 | 7/16 | 3/6 | 2/6 | 4/6 | 7/9 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mg MK-8892-Healthy (N=6) | 1.0 mg MK-8892-Healthy (N=6) | 2.0 mg MK-8892-Healthy (Pooled) (N=6) | 4.0 mg MK-8892-Healthy (N=6) | 6.0 mg MK-8892-Healthy (N=6) | 9.0 mg MK-8892-Healthy (N=6) | 12.0 mg MK-8892-Healthy (N=6) | 14.0 mg MK-8892-Healthy (N=6) | Placebo-Healthy (N=16) | 0.5 mg MK-8892-Hypertensive (N=6) | 1.0 mg MK-8892-Hypertensive (N=6) | 2.0 mg MK-8892-Hypertensive (N=6) | 6.0 mg MK-8892-Hypertensive (N=9) | Placebo-Hypertensive (N=8)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loose stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cyst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Common cold (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Open wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 2 (3) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (with radiation) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 1 (2) | 5 (6) | 4 (4) | 3 (4) | 6 (9) | 4 (6) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 5 (6) | 4 (7)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urtication (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.